CLINICAL TRIAL: NCT05147311
Title: Randomized Trial of a Positive Psychology Intervention for Patients With Hematologic Malignancies Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Positive Psychology Intervention In HSCT
Acronym: PATH-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-362; K08CA251654 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Hematologic Malignancy; Hematopoietic/Lymphoid Cancer; Blood Cancer
Keywords: Hematopoietic Stem Cell Transplant; Positive Psychology; Hematologic Malignancy; Positive Psychological Intervention
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Intervention (Experimental): Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  At approximately 100-days post-HSCT, participants will begin an 9-week positive psychology program involving weekly calls with an interventionist and exercises (i.e., writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  -Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Interventions: Behavioral: Positive Psychology Intervention
- Usual Care Control (No Intervention): Participants in the Usual Care Control arm will receive regular social work assessments as part of HSCT recovery and work does not focus on PPWB skill building or cognitive strategies.

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
  Arms: PATH Intervention

SUMMARY:
The main purpose of this research study is to determine if a positive psychology-based program in people who have received a stem cell transplant for blood cancer treatment is feasible and acceptable, and can help improve positive feelings, mood, quality of life, overall wellbeing and health.

The Positive psychology for Allogenic Transplantation of Hematopoietic stem cell intervention (PATH), a novel 9-week phone-administered Positive psychological intervention (PPI).

DETAILED DESCRIPTION:
Low levels of positive psychological well-being (PPWB) (e.g., optimism, positive affect) in allogeneic hematopoietic stem cell transplant (HSCT) recipients are common and have been associated with decreased quality of life, poorer immune response, and increased mortality. These poor health outcomes are likely mediated through deficits in health behaviors (e.g., medication adherence, physical activity), and indeed low PPWB has been prospectively associated with poorer adherence to diet, medication, and physical activity in other medical populations, independent of sociodemographic, medical comorbidity, and the ill effects of depression and anxiety. Positive psychological interventions (PPIs) could be used to promote PPWB in the allogeneic transplant population. Despite the successful and effective use of PPIs in medical populations to reduce distress, increase quality of life, and promote health behaviors, PPI have never been tested in allogeneic recipients.

-This a single center randomized trial of the PATH intervention versus usual care in patients with hematologic malignancies undergoing HSCT.

The research study procedures include screening for eligibility:

* Participants will be randomized equally to the two arms using randomized permuted blocks of sizes two and four, with randomization stratified by presence/absence of graft-versus-host disease (GVHD), as allogeneic transplant recipients with GVHD have significantly different courses of recovery, QOL, and function post transplant.

  * Participant will be randomized into either: The Positive psychology for Allogenic Transplantation of Hematopoietic stem cell intervention (PATH), a novel 9-week phone-administered Positive psychological intervention (PPI) or usual care.

It is expected that about 70 people will take part in this research study.

The National Institute of Health (NIH), National Cancer Institute (NCI) is supporting this research study by providing funding for the research

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with hematologic malignancies who have received allogeneic HSCT at Dana Farber Cancer Institute who are approaching 100-day post-transplant milestone.
* Ability to speak, read and write English.
* Access to a telephone.

Exclusion Criteria:

* Cognitive deficits impeding a study participant's ability to provide informed consent or participate adequately in the study procedures assessed via a commonly used 6-item cognitive assessment with the Brief Interview for Mental Status (BIMS).
* Medical conditions precluding interviews.
* Patients undergoing HSCT for benign hematologic conditions.
* Patients undergoing outpatient HSCT.
* Patients with psychiatric or cognitive conditions which the treating clinicians believes prohibits compliance with study procedures.
* Patients who are unable to verbally consent or are not yet adults (including infants, children, teenagers), pregnant women, or prisoners.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact study investigator at hermioni_amonoo@dfci.harvard.edu

REFERENCES:
- [Derived] Amonoo HL, Lam JA, Daskalakis E, Deary EC, Celano C, Onyeaka HK, Newcomb R, Barata A, Horick N, Cutler C, Pirl WF, Lee SJ, Huffman JC, El-Jawahri A. Positive Psychological Well-Being in Hematopoietic Stem Cell Transplantation Survivors. Transplant Cell Ther. 2023 Sep;29(9):583.e1-583.e9. doi: 10.1016/j.jtct.2023.07.010. Epub 2023 Jul 11. PMID 37442349

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were not randomized: 1 did not complete baseline measures and 1 was no longer interested in the study.
Groups:
- PATH Intervention: Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  At approximately 100-days post-hematopoietic stem cell transplant (HSCT), participants will begin an 9-week positive psychology program involving weekly calls with an interventionist and exercises (i.e., writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  -Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Positive Psychology Intervention: Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
- Usual Care Control: Participants in the Usual Care Control arm will receive regular social work assessments as part of hematopoietic stem cell transplant (HSCT) recovery and work does not focus on positive psychological well-being (PPWB) skill building or cognitive strategies.
Period: Overall Study
Arm/Group | PATH Intervention | Usual Care Control
Started | 35 | 35
Completed | 31 | 31
Not Completed | 4 | 4
Not completed — Did not complete survey | 2 | 1
Not completed — Patient too sick | 1 | 2
Not completed — Death | 0 | 1
Not completed — Declined survey | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PATH Intervention: Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  At approximately 100-days post-HSCT, participants will begin an 9-week positive psychology program involving weekly calls with an interventionist and exercises (i.e., writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  -Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Positive Psychology Intervention: Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
- Total: Total of all reporting groups
Arm/Group | PATH Intervention | Usual Care Control | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.5) | 56.1 (14.9) | 56.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 13 | 22 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian/Asian background | 3 | 1 | 4
  Race: Black | 1 | 0 | 1
  Race: Native American/Indigenous | 0 | 1 | 1
  Race: White | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Type of cancer [Count of Participants; unit: Participants]
  Leukemia | 23 | 25 | 48
  Lymphoma | 1 | 2 | 3
  Myelodysplastic syndromes/myeloproliferative neoplasms | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Rate
Description: Feasibility was defined a >75% of enrolled participants in the PATH group completing at least 6 of the 9 positive psychology sessions.
Time Frame: 9 weeks
Population: For feasibility analysis based on % of participants who completed ≥6 of 9 sessions sessions, only participants who started the intervention were used. Of the 33 participants who started PATH, 31 (94%) completed ≥6 of 9 sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | PATH Intervention
Number analyzed (Participants) | 33
Participants | 31

2. Secondary Outcome: Acceptability Rate
Description: At the end of each weekly intervention session, acceptability was measured with weekly ratings of ease and utility of each positive psychology exercise with a 10-point Likert scale (0=very difficult/not helpful; 10=very easy/very helpful).
  The mean ease and utility of each exercise was calculated.
Time Frame: 9 weeks
Population: For the acceptability analysis (i.e., mean ease and mean utility analysis), the analysis population denominator was 33 participants in the PATH group. Only participants in the intervention arm provided data on ease and utility since it pertains to the intervention directly.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | PATH Intervention
Number analyzed (Participants) | 33
scores on a scale
  Acceptability - Mean Ease Score | 7.40 [6.87 to 7.92]
  Acceptability - Mean Utility Score | 8.23 [7.83 to 8.63]

3. Secondary Outcome: Mean Quality of Life Scores
Description: 45-item Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) to assess quality of life (QOL) by cohort. Each question is scored from 0 ("Not at all") to 4 ("Very Much"). Total Score range from 0 to 180. A higher score indicates better quality of life. A mean score will be presented for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 99.84 [93.64 to 106.04] | 103.72 [97.52 to 109.92]
  Post-Intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-Intervention (Week 9) | 107.02 [98.96 to 115.08] | 113.82 [105.67 to 121.97]
  Follow-Up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-Up (Week 18) | 111.63 [103.77 to 119.48] | 109.06 [101.10 to 117.02]

4. Other Pre Specified Outcome: Mean Fatigue Score
Description: The Patient Reported Outcome Measurement Information System-Fatigue-8a (PROMIS-Fatigue-8a) questionnaire will be used to assess fatigue by cohort. The total score range is 0-40. A higher score indicates higher levels of fatigue. A mean score will be presented for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 22.26 [19.69 to 24.84] | 21.04 [18.47 to 23.62]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 10.63 [7.87 to 13.39] | 9.36 [6.62 to 12.10]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 10.92 [7.96 to 13.88] | 12.25 [9.18 to 15.31]

5. Other Pre Specified Outcome: Mean Overall Physical Function Score
Description: A mean overall physical function score will be generated for each cohort using a 20-item Patient-Reported Outcomes Measurement Information System-Physical Function-20 (PROMIS-PF-20) with each item scored from 1 to 5. The total score range is 0 to 100. Higher scores indicate better physical function. A mean score will be presented for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 80.11 [77.02 to 83.21] | 84.01 [80.91 to 87.10]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 85.33 [81.32 to 89.33] | 87.07 [83.10 to 91.03]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 87.29 [82.69 to 91.89] | 85.97 [81.26 to 90.69]

6. Other Pre Specified Outcome: Mean Anxiety Score
Description: The 7-item Hospital Anxiety and Depression Scale-Anxiety (HADS-A) was used to assess symptoms of anxiety in all study participants. The total score on the HADS-A subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety or depression. The mean anxiety score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 5.69 [4.50 to 6.88] | 5.20 [4.02 to 6.38]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 3.54 [2.50 to 4.58] | 4.48 [3.45 to 5.51]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 4.27 [3.00 to 5.55] | 5.40 [4.09 to 6.70]

7. Other Pre Specified Outcome: Mean Depression Score
Description: The 7-item Hospital Anxiety and Depression Scale-Depression (HADS-D) was used to assess symptoms of depression. The HADS-D consists of a four-point item response. Scores on the HADS-D subscale range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant depression. The mean depression score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 5.32 [4.26 to 6.37] | 5.02 [3.98 to 6.07]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 4.33 [3.19 to 5.47] | 3.63 [2.50 to 4.75]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 3.91 [2.60 to 5.22] | 4.65 [3.31 to 6.00]

8. Other Pre Specified Outcome: Mean Post-Traumatic Stress Disorder Checklist Score
Description: The 17-item Post-Traumatic Stress Disorder Checklist (PCL) was used to assess symptoms of post-traumatic stress according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders-IV. Each item is scored from 1-5. The total overall score range is 17 to 85. A higher score indicates higher levels of PTSD. A mean score will be presented for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 26.69 [23.80 to 29.58] | 27.27 [24.36 to 30.19]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 25.33 [22.65 to 28.02] | 25.06 [22.38 to 27.74]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 24.31 [21.48 to 27.14] | 27.39 [24.53 to 30.26]

9. Other Pre Specified Outcome: Mean Optimism Score
Description: The 7-item Life Orientation Test-Revised (LOT-R) will be used to measure dispositional (trait) optimism. Each item is scored from 1-5. The total overall score range is 5 to 35. Higher scores indicate greater optimism. A mean score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 17.29 [15.46 to 19.11] | 17.57 [15.75 to 19.40]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 17.99 [16.16 to 19.81] | 18.41 [16.59 to 20.23]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 19.56 [17.84 to 21.27] | 17.14 [15.39 to 18.89]

10. Other Pre Specified Outcome: Mean Positive Affect Score
Description: The 10-item Positive and Negative Affect Schedule (PANAS) will be used to measure positive affect. Each item is scored from 1-5. The total score range is 0 to 50. Higher scores indicate greater positive and negative affect. A mean score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 34.89 [32.42 to 37.36] | 35.54 [33.07 to 38.01]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 36.63 [33.22 to 40.03] | 39.01 [35.57 to 42.45]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 37.82 [34.65 to 40.99] | 36.81 [33.55 to 40.07]

11. Other Pre Specified Outcome: Mean Satisfaction Score
Description: Satisfaction will be measured by Satisfaction with Life Scale (SWLS). This 5 item questionnaire will measure satisfaction with life; higher scores indicate greater satisfaction with life. Each item is scored from 1-7; the total score ranges from 5-35. A mean score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 23.29 [20.81 to 25.76] | 22.65 [20.15 to 25.14]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 22.99 [20.22 to 25.76] | 24.11 [21.32 to 26.91]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 25.16 [22.81 to 27.51] | 23.14 [20.74 to 25.53]

12. Other Pre Specified Outcome: Mean Gratitude Score
Description: The 6-item Gratitude questionnaire (GQ-6) measures dispositional gratitude; higher scores indicate greater proneness to experience gratitude in daily life. Each item will be scored from 1-7; the entire questionnaire will be scored from 6-42. A mean score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 37.51 [36.09 to 38.94] | 37.83 [36.40 to 39.25]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 37.82 [35.90 to 39.75] | 38.03 [36.09 to 39.97]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 38.60 [36.80 to 40.40] | 38.13 [36.29 to 39.96]

13. Other Pre Specified Outcome: Mean Flourishing Score
Description: The 8-item Flourishing Scale measures a person's self-perceived success in critical areas such as engagement, relationships, self-esteem, meaning and purpose, and optimism; higher scores indicate having many psychological resources and strengths. Each item is scored from 1-7; the entire questionnaire is scored from 8-56. A mean score will be reported for each cohort.
Time Frame: At baseline (registration) and then week 9 (+/- 1 week) and week 18 (+/- 1 week) from the time of registration
Population: Intention-to-treat principle was used for all randomized patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PATH Intervention | Usual Care Control
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 51.49 [48.90 to 54.07] | 51.77 [49.19 to 54.35]
  Post-intervention (Week 9): number analyzed (Participants) | 33 | 34
  Post-intervention (Week 9) | 52.02 [48.62 to 55.42] | 55.31 [51.88 to 58.73]
  Follow-up (Week 18): number analyzed (Participants) | 31 | 31
  Follow-up (Week 18) | 52.30 [48.73 to 55.86] | 53.21 [49.59 to 56.84]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the active study period, which lasted from study enrollment through follow-up assessment completion (week 18). Because this was a supportive care intervention, adverse events were not assessed at a pre-specified time. Instead, adverse events were recorded as reported by study participants during the active study period.
Description: This is a population in which disease relapse and death due to transplant complications are to be expected, are not study-related, and were not considered or reported as adverse events for this study. Adverse events related to study procedures were reported to the Institutional Review Board at the PI's discretion. Participants requesting withdrawal from the study were asked to provide reasons for withdrawal to monitor for adverse events or unanticipated events related to study procedures.
Groups:
- PATH Intervention: Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  At approximately 100-days post-HSCT, participants will begin an 9-week positive-psychology program involving weekly calls with an interventionist and exercises (i.e. writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  -Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Positive Psychology Intervention: Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
Arm/Group | PATH Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05147311/Prot_SAP_000.pdf